CLINICAL TRIAL: NCT05456763
Title: Sodium Butyrate Effectiveness in Children and Adolescents With Newly Diagnosed Inflammatory Bowel Diseases - Randomized Placebo-controlled Multicentre Trial
Brief Title: Butyrate in Pediatric Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: nr 41/2013
Record Dates: First submitted 2022-07-06; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Crohn's disease; ulcerative colitis; sodium butyrate
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Butyric Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): 150 mg sodium butyrate twice a day for 12 weeks
  Interventions: Dietary Supplement: sodium butyrate
- group B (Placebo Comparator): placebo capsules twice a day for 12 weeks
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: sodium butyrate — add-on therapy irrespective of standard treatment depending on severity (according to the guidelines)
  Arms: group A
Other: placebo — placebo
  Arms: group B

SUMMARY:
The first prospective randomised placebo-controlled study in the IBD pediatric population was conducted to evaluate the effectiveness of oral sodium butyrate as add-on therapy in IBD.

DETAILED DESCRIPTION:
Butyric acid's effectiveness has not yet been assessed in the pediatric inflammatory bowel disease (IBD) population. This study aimed to evaluate the effectiveness of oral sodium butyrate as an add-on to standard therapy in children and adolescents with newly diagnosed IBD.

This was a prospective, randomized, placebo-controlled multicentre study. Patients aged 6-18 years with colonic Crohn's disease or ulcerative colitis, who received standard therapy depending on the disease's severity, were randomized to receive 150 mg sodium butyrate twice a day (group A) or placebo (group B). The primary outcome was the difference in disease activity and fecal calprotectin concentration between the two study groups measured at 12 weeks of the study.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 18 years of age;
* newly diagnosed, based on the modified Porto criteria, IBD with colon involvement;
* informed consent of the child's parents or guardians to participate in the study.

Exclusion Criteria:

* age <6 years;
* taking probiotics or dietary supplements in the last 2 weeks prior to study enrollment;
* lack of consent of parents or guardians to participate in the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
difference in remission rate (PCDAI for Crohn's disease) | 12 weeks
  The Pediatric Crohn's Disease Activity Index (PCDAI) measured in points of activity was used to assess CD activity.
  Severity of the disease:
  <10 points = remission 10-27.5 points = mild Crohn's Disease 30-37.5 points = moderate Crohn's Disease
  ≥40 points = severe Crohn's Disease
  In this scale addominal pain (mild or moderate/severe), number of stools per day, general well being (good, below par, very poor), antropometric measures, palpable mass in the abdomen and perianal fistulas are assessed. The scale is validated and used in daily clinical practice.
  Remission was defined as less than 10 points for both PCDAI and PUCAI scores.
difference in remission rate (PUCAI ulcerative colitis) | 12 weeks
  The Pediatric Ulcerative Colitis Activity Index (PUCAI) measured in points of activity was used to assess UC activity.
  Severity of the disease:
  <10 points = remission 10-34 points = mild ulcerative colitis 35-64 points = moderate ulcerative colitis
  ≥65 points = severe ulcerative colitis
  In this scale addominal pain (mild or moderate/severe), number of stools per day, blood in the stool, stool consistency, nocturnal stools and activity level (no limitation, occasional or restricted), are assessed. The scale is validated and used in daily clinical practice.
  Remission was defined as less than 10 points for both PCDAI and PUCAI scores.

SECONDARY OUTCOMES:
difference in disease activity for CD and UC patients | 12 weeks
  assessed separately, calcultated in points (described above)
difference in calprotectin concentration | 12 weeks
  measured in µg/g assessed in different soubgroups (lower result is better, remission = less than 50.
side effects | 12 weeks
  assessed for both groups (descriptive)